CLINICAL TRIAL: NCT06738225
Title: Serum MicroRNAs as Diagnostic Biomarkers of Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Bishoy Shehata (Other)
Responsible Party: Sponsor-Investigator, Bishoy Shehata, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: MicroRNAs , colorectal cancer
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: MicroRNAs; Colorectal Cancer; miR-15b; miR-21
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Persons has Colorectal cancer
  Interventions: Diagnostic Test: certain serum MicroRNA biomarkers (miR-15b and miR-21)
- Control: Persons do not have Colorectal cancer
  Interventions: Diagnostic Test: certain serum MicroRNA biomarkers (miR-15b and miR-21)

INTERVENTIONS:
Diagnostic Test: certain serum MicroRNA biomarkers (miR-15b and miR-21) — miR-15b and miR-21 as diagnostic biomarkers of colorectal cancer

SUMMARY:
evaluation the diagnostic value of certain MicroRNAs as biomarkers of Colorectal cancer by comparing its expression levels in Colorectal cancer patients and normal individuals.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second commonest cause of cancer deaths and the third most common cancer worldwide. Five year survival of patients with stage 1 CRC is 92%, and decreases to 10% at stage 4 CRC. So, CRC diagnosing at an early stage is the most important factor influencing disease prognosis. Most CRC patients are diagnosed after being symptomatic, but studies show that once the symptoms are present it mostly signifies late-stage disease. colonoscopic screening of asymptomatic patients has been shown to pick up early-stage CRC. However, this is limited by cost issues and patient attitudes. Therefore, more efforts could be done to view to early diagnosis of CRC in asymptomatic patient. Biomarkers are molecules that can serve as signals of disease activity and pathological processes. CRC biomarkers can help in early diagnosis. MicroRNAs (miRNAs) are non-coding molecules that impact the expression of target genes in cell. Also, they exist in highly stable, cell free form in peripheral blood. They are detected by quantitative real time polymerase chain reaction (qRT-PCR). Data also shows that certain miRNAs are elevated in the plasma and tissues of CRC patients and decrease in plasma levels after operative treatment. There are over 2000 different miRNAs and they are estimated to regulate 30% of the human genome. miRNA dysregulation is also associated with multiple cancers. miRNAs seem to show significant promise with high sensitivity and specificity for CRC, but with limiting factors of limited data for high risk polyps and significant heterogeneity in test media and non-standardisation of test panels. Further research would be required to bridge these knowledge gaps. Interestingly, miR-15b and miR-21 appears to be the best diagnostic accuracy values for CRC.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-75) diagnosed with primary CRC (histopathologically confirmed).
* CRC patients who have not received prior treatment (i.e., chemotherapy or radiation).
* Age-matched healthy controls without colorectal disease

Exclusion Criteria:

* Patients with secondary tumors or metastasis originating from non-colorectal sources.
* Patients with prior history of CRC.
* Patients who refuse to contribute in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
evaluation the diagnostic value of miRNAs as biomarkers of CRC by comparing its expression levels in CRC patients and normal individuals | baseline
  use the results of measurement of certain serum miRNAs in persons with CRC and non-CRC individuals.

SECONDARY OUTCOMES:
assessment the correlation between miRNAs expression levels and clinicopathological features such as tumor stage, grade, and metastasis | baseline
  use the results of measurement of certain serum miRNAs in persons with CRC and non-CRC individuals.
evaluation the sensitivity, specificity, and diagnostic accuracy of miRNAs as standalone biomarkers | baseline
  use the results of measurement of certain serum miRNAs in persons with CRC and non-CRC individuals.

IPD SHARING:
Plan to Share IPD: No